CLINICAL TRIAL: NCT00569530
Title: Trial of Late Surfactant to Prevent BPD: A Pilot Study in Ventilated Preterm Neonates Receiving Inhaled Nitric Oxide
Acronym: TOLSURFPilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Roberta Ballard (Other)
Collaborators: Mallinckrodt (Industry); ONY (Industry)
Responsible Party: Sponsor-Investigator, Roberta Ballard, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H10842-31630-01; IND79367 (Other: FDA)
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Distress Syndrome of Prematurity (Surfactant Dysfunction); Bronchopulmonary Dysplasia
Keywords: nitric oxide; surfactant; bronchopulmonary dysplasia; prematurity; neonates; iNO; Infasurf; lung function; ventilated infants
MeSH Terms: conditions — Respiratory Distress Syndrome; Surfactant Dysfunction; Bronchopulmonary Dysplasia; Premature Birth | interventions — calfactant; salicylhydroxamic acid; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Surfactant (Infasurf) ONY, NY (Active Comparator): Patients receive inhaled nitric oxide and scheduled doses of Infasurf on study days 0, 3, 7, 10, and 14, if infant remains ventilated.
  Interventions: Drug: Infasurf (ONY Inc.)
- Sham (no treatment) (Placebo Comparator): Infants receiving inhaled nitric oxide will receive Sham (no treatment) on study days 0, 3, 7, 10, and 14, if infant remains ventilated.
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Infasurf (ONY Inc.) — Infasurf 3ml/kg will be given to infants on study days 0, 3, 7, 10, and 14, if remains intubated.
  Other Names: Infasurf
  Arms: Treatment Surfactant (Infasurf) ONY, NY
Drug: Sham — Sham instillation (no treatment) will be given to study infants on days 0, 3, 7, 10, and 14, if remains intubated.
  Other Names: Air
  Arms: Sham (no treatment)

SUMMARY:
The purpose of this study is to determine if the combination of late doses of Infasurf with inhaled nitric oxide will interact to improve the surfactant function and thus the respiratory status and outcome of treated infants.

DETAILED DESCRIPTION:
Surfactant dysfunction may contribute to the development of bronchopulmonary dysplasia (BPD) in persistently ventilated preterm infants. The investigators conducted a multi-center, randomized, blinded pilot study to assess the safety and efficacy of late administration of surfactant (Calfactant - high in protein B) in combination with prolonged inhaled nitric oxide in preterm infants < 1000 grams birthweight (BW). Calfactant is one of several types of exogenous surfactant. Calfactant has the highest % of surfactant protein B of the different types.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 1000 gm. birth weight
* Less than or equal to 30 weeks gestational age
* Day 7-14 of life
* Intubated and mechanically ventilated at any time days 7-14 of life

Exclusion Criteria:

* Serious congenital malformations
* Life expectancy less than 7 days from enrollment
* Previous treatment with iNO
* Active pulmonary hemorrhage at time of enrollment
* Active air leak syndrome at time of enrollment
* Bilateral grade IV intracranial hemorrhage prior to enrollment
* Less than 48 hours from last clinical dose of early surfactant.

Ages: 7 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A Ballard, MD, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - Alta Bates Summit Medical Center, Berkeley, California
  - Children's Hospital Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Mercy Hospital, Kansas City, Missouri
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballard RA, Truog WE, Cnaan A, Martin RJ, Ballard PL, Merrill JD, Walsh MC, Durand DJ, Mayock DE, Eichenwald EC, Null DR, Hudak ML, Puri AR, Golombek SG, Courtney SE, Stewart DL, Welty SE, Phibbs RH, Hibbs AM, Luan X, Wadlinger SR, Asselin JM, Coburn CE; NO CLD Study Group. Inhaled nitric oxide in preterm infants undergoing mechanical ventilation. N Engl J Med. 2006 Jul 27;355(4):343-53. doi: 10.1056/NEJMoa061088. PMID 16870913
- [Background] Ballard PL, Merrill JD, Truog WE, Godinez RI, Godinez MH, McDevitt TM, Ning Y, Golombek SG, Parton LA, Luan X, Cnaan A, Ballard RA. Surfactant function and composition in premature infants treated with inhaled nitric oxide. Pediatrics. 2007 Aug;120(2):346-53. doi: 10.1542/peds.2007-0095. PMID 17671061
- [Background] Truog WE, Ballard PL, Norberg M, Golombek S, Savani RC, Merrill JD, Parton LA, Cnaan A, Luan X, Ballard RA; Nitric Oxide (to Prevent) Chronic Lung Disease Study Investigators. Inflammatory markers and mediators in tracheal fluid of premature infants treated with inhaled nitric oxide. Pediatrics. 2007 Apr;119(4):670-8. doi: 10.1542/peds.2006-2683. PMID 17403837
- [Background] Keller RL, Merrill JD, Black DM, Steinhorn RH, Eichenwald EC, Durand DJ, Ryan RM, Truog WE, Courtney SE, Ballard PL, Ballard RA. Late administration of surfactant replacement therapy increases surfactant protein-B content: a randomized pilot study. Pediatr Res. 2012 Dec;72(6):613-9. doi: 10.1038/pr.2012.136. Epub 2012 Oct 4. PMID 23037875

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Surfactant (Infasurf) ONY, NY: Patients receive inhaled nitric oxide and scheduled doses of Infasurf on study days 0, 3, 7, 10, and 14, if infant remains ventilated.
  Infasurf (ONY Inc.): Infasurf 3ml/kg will be given to infants on study days 0, 3, 7, 10, and 14.
- Sham (no Treatment): Infants receiving inhaled nitric oxide will receive Sham (no treatment) on study days 0, 3, 7, 10, and 14, if infant remains ventilated.
  Sham Infants will not receive additional doses of Infasurf.
Period: Overall Study
Arm/Group | Treatment Surfactant (Infasurf) ONY, NY | Sham (no Treatment)
Started | 43 | 42
Completed | 43 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Surfactant (Infasurf) ONY, NY | Sham (no Treatment) | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: Days] — Age at enrollment: Infants were enrolled if they remained ventilated between 7 and 14 day of age.
  Days | 9.9 (2.2) | 10.5 (2.8) | 10.2 (2.5)
Sex/Gender, Customized [Number; unit: infants]
  Female | 14 | 23 | 37
  Male | 29 | 19 | 48
Race/Ethnicity, Customized [Number; unit: infants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 25 | 32 | 57
  Unknown or Not Reported | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: infants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 16 | 25
  White | 29 | 24 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: infants]
  United States | 43 | 42 | 85
Antenatal Corticosteroids [Number; unit: infants] — Number of infants who received Antenatal Corticosteroids. Not all mothers receive antenatal steroids. Therefore number treated will not match number in group.
  infants | 32 | 33 | 65
Prior surfactant treatment [Number; unit: infants] — Number of infants who received prior surfactant therapy (prior to enrollment). Not all infants receive surfactant therapy at birth. Therefore number treated will not always match number in group.
  infants | 43 | 41 | 84
RSS at entry [Mean (Standard Deviation); unit: cm H2O] — Respiratory Severity Score = Mean Airway pressure X FiO2. The higher the number, the sicker the infant.
  cm H2O | 3.4 (1.7) | 3.2 (1.7) | 3.3 (1.7)
Multiple gestation [Number; unit: infants] — The number of infants who were a product of a multiple gestation pregnancy. Only a small number of pregnancies are multiple gestation. Multiple gestation infants will be a subset of infants enrolled.
  infants | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: SP-B Content
Description: SP-B Content is the surfactant protein B found in terms of percentage of phospholipid measured one day after surfactant or sham dose.
Time Frame: One day after dose
Population: 24 of 43 in the Treatment Group and 18 of 42 in the Sham group had samples analyzed. SpB content recorded as a percentage of Total Phospholipids.
Measure: Mean (Full Range); unit: Total surfactant protein (% of PL)
Arm/Group | Treatment Surfactant (Infasurf) ONY, NY | Sham (no Treatment)
Number analyzed (Participants) | 24 | 18
Total surfactant protein (% of PL) | 19.9 [3.7 to 71.0] | 13.3 [4.3 to 47.8]

2. Secondary Outcome: Alive Without BPD at 36 Weeks Post Menstrual Age
Description: Alive without need for oxygen at 36 weeks post menstrual age.
Time Frame: 36 Weeks Post Menstrual Age
Measure: Number; unit: Number of infants
Arm/Group | Treatment Surfactant (Infasurf) ONY, NY | Sham (no Treatment)
Number analyzed (Participants) | 43 | 42
Number of infants | 16 | 14

ADVERSE EVENTS:
Arm/Group | Treatment Surfactant (Infasurf) ONY, NY | Sham (no Treatment)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

LIMITATIONS AND CAVEATS:
More frequent dosing, with the resultant improvements in lung function, may allow for more rapid weaning from mechanical ventilation, leading to improved pulmonary outcomes, both short-term and long-term. Modifications to protocol being investigated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No